CLINICAL TRIAL: NCT01796158
Title: Pilot Test of Computerized MET Intervention to Reduce Adolescent Alcohol Use
Brief Title: Pilot Test of Computerized MET to Reduce Adolescent Alcohol Use
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not funded
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JKR34_PA-13-078
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Abuse
Keywords: adolescents; alcohol abuse; drug abuse; substance use
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cASBI+cMET (Experimental): Participants will complete the computerized alcohol screening and brief intervention (cASBI)protocol at the time of an office visit and also complete the 2-session computerized Motivational Enhancement Therapy intervention (cMET).
  Interventions: Behavioral: cASBI+cMET; Behavioral: cASBI
- cASBI (Active Comparator): Participants will complete the computerized screening and brief intervention protocol at the time of a primary care office visit.
  Interventions: Behavioral: cASBI

INTERVENTIONS:
Behavioral: cASBI+cMET — In the cASBI protocol participants complete a computerized screen for alcohol and drug use, view their screen results on the computer, then see 10 pages of science and true life stories describing the health effects of alcohol and other substance use. The provider receives a report of the screen results and gives brief advice regarding alcohol and drug use during the office visit. The cMET protocol is a 2 session intervention composed of 8 exercises designed to encourage adolescents their alcohol and other substance use and develop a plan to stop or reduce their use.
  Arms: cASBI+cMET
Behavioral: cASBI — In the cASBI protocol participants complete a computerized screen for alcohol and drug use, view their screen results on the computer, then see 10 pages of science and true life stories describing the health effects of alcohol and other substance use. The provider receives a report of the screen results and gives brief advice regarding alcohol and drug use during the office visit.

SUMMARY:
The goal of this project is to conduct a pilot study evaluating feasibility, acceptability, and estimating the effect size of a new computerized Motivational Enhancement Therapy (cMET) intervention for alcohol-involved adolescent primary care patients.

DETAILED DESCRIPTION:
The goal of this project is to conduct a pilot study evaluating feasibility, acceptability, and estimating the effect size of a new computerized Motivational Enhancement Therapy (cMET) intervention for alcohol-involved adolescent primary care patients. The investigators hypothesize that 1) cMET, when added to Computerized Alcohol Screening and Brief Intervention (cASBI), (cASBI+cMET) will be feasible and acceptable when used in primary care; and 2) 12- to 18-yr old patients receiving cASBI+cMET will have lower rates of any alcohol use, days of alcohol use, drinks per drinking day, and days of heavy episodic drinking, than cASBI alone.

ELIGIBILITY:
Inclusion Criteria:

* any alcohol use days in the past 90 days
* have an email address and internet access at home, school, or library

Exclusion Criteria:

* unable to read or understand English
* living away at college at the time of the recruitment visit
* not available for computer/telephone follow-ups
* judged by the provider to be medically or emotionally unstable at time of visit

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
cMET completion | Baseline
  The investigators will measure the percentages of completed cMET sessions by those referred to cMET.

SECONDARY OUTCOMES:
cMET satisfaction | 9 months
  The investigators will measure patient satisfaction with the cMET program.

OTHER OUTCOMES:
Alcohol use | 9 months
  The investigators will measure rates of any alcohol use, days of alcohol use, drinks per drinking day, and days of heavy episodic drinking in the cASBI+cMET group vs the cASBI group.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No